CLINICAL TRIAL: NCT07089459
Title: Low Level Laser Therapy Versus Short Wave Diathermy in Patients With Anterior Cruciate Ligament Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sana Ali, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/505/08/24
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear
Keywords: Functional Disability; Knee Pain; Low-Level Laser Therapy; Muscle Strength; Photobiomodulation; Short wave therapy
MeSH Terms: conditions — Lacerations | interventions — Low-Level Light Therapy; Short-Wave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Level Laser Therapy (Experimental): Participants in this arm will receive Low-Level Laser Therapy (LLLT) along with standard physiotherapy exercises and shortwave diathermy. LLLT will be administered 2-3 times per week for 6 weeks using an 830 nm wavelength, 150 mW power output, and 5 W/cm² power density. Standard exercises include heel slides, partial knee bends, quad sets, and step-ups. Shortwave diathermy will be delivered at 27.12 MHz frequency, 20-30 minutes per session. The intervention aims to improve pain, strength, and functional disability in patients with partial ACL tears.
  Interventions: Device: Low-Level Laser Therapy (LLLT)
- Shortwave therapy (Active Comparator): Participants in this arm will receive standard physiotherapy combined with shortwave diathermy (SWD), without the addition of Low-Level Laser Therapy (LLLT). The physiotherapy protocol includes supervised exercises such as heel slides, partial knee bends, quadriceps sets, and step-ups. SWD will be administered 2-3 times using a 27.12 MHz frequency for 20-30 minutes per session. This arm serves as the control group to evaluate the added clinical value of LLLT in the conservative management of partial ACL tears.
  Interventions: Behavioral: Shortwave therapy

INTERVENTIONS:
Device: Low-Level Laser Therapy (LLLT) — Low-Level Laser Therapy (LLLT) will be administered using an 830 nm wavelength and 150 mW power output with 5 W/cm² power density. The laser probe will be applied 2-3 times per week for 6 weeks over the affected knee. Treatment is performed using a direct skin contact method with 3-4 minutes of exposure per point around the knee joint. The goal is to reduce inflammation, enhance collagen synthesis, and support ligament healing in patients with partial anterior cruciate ligament (ACL) tears. This intervention is provided in addition to standard physiotherapy and shortwave diathermy.
  Arms: Low-Level Laser Therapy
Behavioral: Shortwave therapy — Participants in this group will receive standard physiotherapy exercises combined with shortwave diathermy (SWD), without the application of Low-Level Laser Therapy (LLLT). The exercise protocol includes heel slides, supported partial knee bends, quadriceps sets, and step-ups, performed in 2 sets of 10 repetitions with 3-5 second rest intervals. SWD will be delivered 2-3 times, using a 27.12 MHz frequency for 20-30 minutes per session, targeting pain relief and enhanced soft tissue healing. This group functions as an active comparator to assess the additional therapeutic value of LLLT used in the intervention group.
  Arms: Shortwave therapy

SUMMARY:
This clinical research study is comparing two non-surgical treatments-Low-Level Laser Therapy (LLLT) and Short Wave Diathermy (SWD)-to see which is more effective for people with a partial tear of the anterior cruciate ligament (ACL) in the knee. The ACL is a key ligament that helps keep the knee stable during movement. When partially torn, it can cause pain, weakness, and difficulty with walking or physical activities.

LLLT, also called photobiomodulation, is a painless, light-based therapy that helps reduce swelling, relieve pain, and promote healing. SWD is a type of deep heat therapy commonly used in physiotherapy to improve circulation and tissue repair.

This study will include 72 patients between 20 and 40 years old who have been diagnosed with a partial ACL tear through MRI. All participants will receive standard physiotherapy exercises and SWD, while half will also receive LLLT.

The study aims to find out if adding LLLT can:

Reduce knee pain

Improve knee muscle strength

Help patients perform daily activities more easily

Each participant will be monitored for 6 weeks, with check-ins at the start, the 3rd week, and the 6th week. Pain levels, muscle strength, and knee function will be measured using reliable assessment tools. The results of this study may help guide better treatment options for people with ACL injuries who want to avoid surgery.

DETAILED DESCRIPTION:
Background & Rationale:

Partial anterior cruciate ligament (ACL) tears are frequent orthopedic injuries, particularly among young adults involved in sports requiring rapid pivoting or directional changes. These injuries often result in pain, instability, muscular weakness, and functional limitations. While complete ACL tears often necessitate surgical reconstruction, partial tears are typically managed with conservative approaches such as physiotherapy and adjunctive non-invasive therapies.

Low-Level Laser Therapy (LLLT), or photobiomodulation, is a non-thermal modality that promotes tissue healing through light-induced cellular stimulation. It has shown beneficial effects in reducing inflammation and pain across various musculoskeletal conditions. However, there is limited high-quality evidence evaluating its specific effects on partial ACL injuries or how it compares to widely used modalities like Short Wave Diathermy (SWD).

Study Design and Methodology:

This is a single-blinded, randomized controlled trial enrolling 72 participants aged 20-40 years with MRI-confirmed partial ACL tears. Participants are randomly assigned (n=36 each) into two groups:

Group A (LLLT + SWD + Physiotherapy): Receives Low-Level Laser Therapy in addition to standard physiotherapy and short wave diathermy

Group B (SWD + Physiotherapy): Receives standard physiotherapy and short wave diathermy only

LLLT Protocol:

Wavelength: 830 nm

Power Output: 150 mW

Power Density: 5 W/cm²

Frequency: 2-3 sessions per week for 6 weeks

Application Time: 3-4 minutes per treatment site (targeting multiple anatomical points around the knee)

Standard Physiotherapy for Both Groups:

Exercises: Heel slides, partial knee bends, quadriceps sets, step-ups

Repetitions: 2 sets of 10, with 3-5 second rest intervals

Short Wave Diathermy Protocol (Both Groups):

Frequency: 27.12 MHz

Duration: 20-30 minutes per session

Application: 2-3 sessions over baseline phase

Outcome Measures:

Assessments will be conducted at baseline, 3rd week, and 6th week using validated clinical tools:

Pain: McGill Pain Questionnaire

Muscle Strength: Handheld dynamometer (quadriceps/hamstrings)

Functional Disability: KOOS (Knee Injury and Osteoarthritis Outcome Score)

Blinding and Randomization:

Random allocation via computerized random number generation

Single-blinded: Outcome assessors blinded to group assignment

Ethical Approval and Consent:

Approved by the Ethical Review Committee at the University of Lahore

Informed written consent obtained from all participants

Privacy and confidentiality strictly maintained

Expected Impact:

This study aims to provide evidence on whether LLLT offers superior clinical outcomes in pain relief, strength enhancement, and functional recovery compared to SWD in the conservative management of partial ACL injuries. The findings may help refine treatment protocols, promote cost-effective and non-invasive rehabilitation options, and guide physiotherapists in evidence-based practice.

ELIGIBILITY:
Inclusion Criteria:

* Pain in knee lasting more than 15 days (Masiero et al., 2020)
* Unilateral partial ACL tear diagnosed with positive lachman test and negative pivot shift test (+ve pivot shift leads to complete tear) with or without other ligament tear (Song et al., 2024)
* No other osteoarticular or soft tissue lesion (Masiero et al., 2020)

Exclusion Criteria:

* Patients with tumors or other serious diseases (Song et al., 2024)
* History of deep vein thrombosis or vascular pathology in any lower limb (Song et al., 2024)
* Rheumatoid arthritis or other signifcant co-morbidities (Masiero et al., 2020)
* Intraarticular injections into the knee in the preceding 6 months (Song et al., 2024)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Functional Disability Assessed by KOOS | Baseline, 3rd week, and 6th week
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) will be used to evaluate functional disability in participants with partial ACL tears. KOOS is a validated, 42-item questionnaire assessing five subscales: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. Higher scores indicate better knee function and less disability. The score will be compared between groups over time to determine the effectiveness of LLLT in improving knee function.

SECONDARY OUTCOMES:
Change in Pain Intensity Assessed by McGill Pain Questionnaire | Baseline, 3rd week, and 6th week
  Pain intensity will be measured using the McGill Pain Questionnaire, a multidimensional tool that assesses sensory, affective, and evaluative aspects of pain through 78 descriptors. The total pain rating index will be calculated based on participant responses. A reduction in the score will indicate decreased pain severity.
Change in Knee Muscle Strength Measured by Handheld Dynamometer | Baseline, 3rd week, and 6th week
  Knee extensor and flexor muscle strength will be assessed using a handheld dynamometer. Participants will perform isometric contractions while force output is measured in Newtons. Improvements in strength values over time will indicate muscular recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masiero S, Pignataro A, Piran G, Duso M, Mimche P, Ermani M, Del Felice A. Short-wave diathermy in the clinical management of musculoskeletal disorders: a pilot observational study. Int J Biometeorol. 2020 Jun;64(6):981-988. doi: 10.1007/s00484-019-01806-x. Epub 2019 Nov 20. PMID 31748973